CLINICAL TRIAL: NCT03672500
Title: Analgesic Benefit of Locally Injected Bupivacaine on Perineal Pain Among Women With Epidural Anesthesia After a Vaginal Delivery: a Randomized, Single-masked, Controlled Trial
Brief Title: Perineal Local Infiltration Study
Acronym: PLIS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment issues
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: PLIS_1
Record Dates: First submitted 2018-03-26; First posted 2018-09-14 (Actual); Last update posted 2022-05-18 (Actual); Status verified 2022-05

CONDITIONS: Second Degree Perineal Tear During Delivery - Delivered; Episiotomy; Complications; Anesthesia, Local
MeSH Terms: interventions — Bupivacaine; salicylhydroxamic acid

STUDY DESIGN:
Intervention Model Description: a randomized, single-masked, controlled trial
Who Masked: Participant, Outcomes Assessor
Masking Description: a randomized, single-masked, controlled trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bupivacaine arm (Active Comparator): The edges of the 2PT/Epi will be infiltrated with 10ml of Bupivacaine 0.5%+Epinephrine 50mcg prior to suture placement.
  Interventions: Drug: Bupivacaine 0.5%+Epinephrine 50mc
- Control arm (Sham Comparator): Sham injection will be done using a syringe filled with 10ml of NaCl 0.9%, but the fluid will not be injected to the edges of the laceration but discarded. The sham injection will last no less than 10 seconds.
  Interventions: Other: Sham injection

INTERVENTIONS:
Drug: Bupivacaine 0.5%+Epinephrine 50mc — Local infiltration of the perineum with Bupivacaine 0.5%+Epinephrine 50mc
  Arms: Bupivacaine arm
Other: Sham injection — Sham injection of the perineum
  Arms: Control arm

SUMMARY:
The prevalence of birth canal lacerations is more than 70% of all deliveries in Canada. The repair of such lacerations is usually done using a pre-existing epidural analgesia. Once the analgesic effect of the epidural analgesia fades, the laceration may cause intolerable pain, and result in emotional stress, difficulties in ambulation and breastfeeding, and more.

The research team hypothesis is that adding a locally injected analgesic, which will take effect once the epidural analgesia fades, may alleviate perineal pain, prevent such difficulties, and improve women's overall well-being and satisfaction.

The proposed trial is a two-arm, single-masked, randomized trial. Women with a working epidural analgesia, and a laceration will be invited to participate. Women in the local anesthesia (LA) arm will get a LA injected to the laceration and women in the sham arm will get no injection. The differences in perineal pain between the groups will be evaluated at 6 hours after last epidural dose.

DETAILED DESCRIPTION:
1. The Need for the Trial

   1.1. Background

   Perineal trauma during delivery may be iatrogenic (episiotomy) or spontaneous (perineal tear). First-degree injury involves the perineal skin only, while a 2nd-degree perineal tear (2PT) involves perineal muscles as well1,2. A 3rd-degree tear involves the anal sphincter, and a 4th-degree tear involves the entire anal sphincter complex (external and internal anal sphincters) and the anal epithelium1,2. An episiotomy (Epi) is usually performed in a mediolateral or lateral manner, and is considered a 2nd degree laceration by definition. The morbidity associated with obstetrical anal sphincter injury (3rd or 4th degree perineal tear) is considerably higher than in 1st or 2nd degree tear1,2.

   The repair of a perineal tear may be done using the epidural anesthesia that was used during delivery, with no additional analgesia. If the patient is delivered without an epidural anesthesia, a short-acting local anesthetic agent, such as lidocaine, may be infiltrated to the edges of the wound prior to suturing.

   Scope of the problem The annual number of deliveries in Canada approaches 390,000, of which more than 145,000 are anticipated to take place in Ontario3. It has been reported that approximately 70% of deliveries in Ontario are vaginal deliveries4. Episiotomies occur in approximately 20% of vaginal deliveries, with 50% a 1st or 2nd degree perineal tear occur, and 3.2% of vaginal deliveries are complicated by a 3rd or 4th degree perineal tear4,5.

   Pain and morbidity associated with perineal lacerations Numerous studies have addressed the short- and long-term pain and morbidity associated with perineal lacerations. While numbers vary according to local practices and cultural and ethnical differences, most agree that perineal trauma is a major source of pain and morbidity6-12. Most studies reported Numeric Rating Scale (NRS) or Visual Analog Scale (VAS) scores in which pain is ranked by the patient verbally (from 0 to 10) or on a 10-cm ruler13, respectively. Some of the studies have reported VAS scores associated with 2PT/Epi of more than 5, and up to 8.5, in the first postpartum day7,9,12. Moreover, it has been shown that perineal lacerations, iatrogenic or spontaneous, are associated with interference with daily activities such as sitting, ambulation, urination and bowel movements14-19. Some have reported that more than 55% of women with 2PT/Epi experienced interference with at least one daily activity that was attributed to perineal pain7, and others have shown that between 45-75% of women with 2PT/Epi complained of at least moderate pain while sitting or moving10. Perineal pain associated with 2PT/Epi was also found to interfere with breastfeeding, and proper analgesia was found to have a beneficial effect on this matter14-16. Furthermore, acute pain during the immediate postpartum period was found to be associated with a higher risk of persistent pain 8 weeks postpartum, as well as with the development of postpartum depression7. The authors hypothesized that the severity of acute pain is not just a marker for the development of persistent pain, but also plays a role in the plasticity pathophysiology of acute-to-chronic pain transition.

   Pain relief - current practice

   As stated, perineal tear is usually repaired and sutured using the pre-existing epidural anesthesia that was used for delivery. Once the epidural anesthesia fades, the women will likely experience some perineal pain, mainly during the first 24 hours postpartum. Several studies have examined the benefits of different analgesic regimens, including oral or rectal analgesics, non-pharmacological methods, and topical anesthetics20-25. In most institutions, oral analgesics are provided, whether in a pre-scheduled analgesic plan or as per patient request.

   Despite efforts to alleviate perineal pain, current acceptable pain management protocols have several limitations. First, the use of systematic medications in order to treat local pain may induce side effects, and fail to target the specific pain on the other. Second, many women have concerns regarding the use of systemic medications along with breastfeeding, despite reassurance from medical staff. Topically applied anesthetics were not proven to alleviate postpartum perineal tear, and rectal analgesia was only studied as a single agent compared to placebo, and not as an adjunct to commonly used pain management protocols, thus no superiority was shown.

   At Sunnybrook Health Sciences Centre), a per-patient-request protocol is instituted, which includes acetaminophen (oral, 1000mg every 6 hours, PRN) and naproxen (oral, 400mg every 6 hours, PRN). Additionally, patients may ask for topical lidocaine 4% solution and oral oxycodone 5-10 mg every 4 hours (up to 40 mg/day in breastfeeding mothers).

   1.2. Hypothesis

   Injecting a long-acting local anesthetic into the edges of 2PT/Epi, before suturing, in women who had a vaginal delivery with an epidural anesthesia, will provide longer and more efficient pain relief compared with the common practice of not using local anesthetics.

   1.3. Research questions

   1.3.1. Primary research question

   Using the PICOT technique, the primary research question addresses five main aspects of the trial: population, intervention, comparison, outcome, and time.

   P: In women who have had a vaginal delivery under an epidural anesthesia and have experienced an episiotomy or a 2nd degree perineal tear, I: Does the local injection of bupivacaine to the edges of 2PT/Epi C: compared to a current practice of no analgesic O: increase or decrease perineal pain T: 6 hours after last epidural bolus?

   1.3.2. Other research questions

   In women who have had a vaginal delivery under an epidural anesthesia and have experienced an episiotomy or a 2nd degree tear, does the local injection of bupivacaine to the edges of 2PT/Epi compared to no analgesic increase or decrease -
   * Time to first ambulation (getting out of bed for any activity).
   * Time to first analgesic administration.
   * Number of analgesics administrations during the 24 hours after last epidural bolus.
   * Perineal pain at 12 and 24 hours (±30 minutes) after last epidural bolus.
   * Most severe perineal pain in rest during the first 12 and 24 hours after last epidural bolus.
   * Most severe perineal pain while sitting during the first 12 and 24 hours after last epidural bolus.
   * Most severe perineal pain during walking and breastfeeding during the first 12 and 24 hours after last epidural bolus.
   * Most severe perineal pain during breastfeeding during the first 12 and 24 hours after last epidural bolus.
   * Most severe perineal pain in rest, sitting, walking and breastfeeding during the first 12 and 24 hours after last epidural bolus.

   1.4. Supporting evidence for the hypothesis

   Potential intervention - local infiltration of surgical wound with local anesthetics

   Local anesthetics have been used in multimodal anesthesia regimens in order to reduce the need for post-operative analgesia, mainly opioids26. Several reports have demonstrated the efficacy of local infiltration of anesthetics in surgical wounds. Some have found reductions in both post-operative analgesia use and VAS scores, while some reported more modest outcomes27-33.

   Local infiltration of perineal lacerations with local anesthesia agent or saline

   Two studies have examined infiltration of perineal laceration as a preventative measure to provide longer-acting pain relief once the epidural anesthesia fades.

   The first, by Khan and Lilford, dates back to 198734. In their study, they compared three groups of women with episiotomies (50 women in each group): group 1 had an epidural anesthesia, group 2 had an epidural anesthesia and local infiltration of saline, and group 3 did not have epidural anesthesia, and received lignocaine prior to suture of the episiotomy. They excluded women with large perineal tears, extended episiotomies or third degree perineal tears. They have found that both group 2 and 3 had lower pain scores on day 1 postpartum, and that group 2 (epidural + saline) had the lowest pain scores. They concluded that the artificial swelling induced by the infiltrated agents (regardless of which agent) accommodates the inflammatory edematous response, thus preventing the compression of the tissue by the sutures, and preventing the pain resulting from it. This study had some limitations in that it was not blinded, it excluded perineal tears, was performed three decades ago when practices were different, and did not control for different confounders.

   The second report is more recent, yet only patients with episiotomies were included35. In this double-blind randomized prospective study, infiltration with 15 mL of 0.75% ropivacaine, 1% lidocaine, or saline was performed immediately before initiating the perineal repair. A total of 154 patients were included. The authors did not find any differences between time to first oral analgesic request or pain scores during the first 24 hours postpartum. Yet, while this study employed a more adequate methodology, it did not compare patients to common practice (which is to infiltrate no agent), it included only women with episiotomies and excluded women with operative vaginal deliveries, and did not report the power of the study.

   Bupivacaine

   Bupivacaine Hydrochloride is 2-Piperidinecarboxamide, 1-butyl-N-(2,6-dimethylphenyl)-monohydrochloride, monohydrate, a white crystalline powder that is freely soluble in 95 percent ethanol, soluble in water, and slightly soluble in chloroform or acetone. It is available in sterile isotonic solutions with and without epinephrine (as bitartrate) 1:200,000 for injection via local infiltration, peripheral nerve block, and caudal and lumbar epidural blocks. It is related chemically and pharmacologically to the aminoacyl local anesthetics, and is chemically related to lidocaine.

   The onset of action with Bupivacaine Hydrochloride is rapid and anesthesia is long lasting. The duration of anesthesia is significantly longer with Bupivacaine Hydrochloride than with any other commonly used local anesthetic. It has also been noted that there is a period of analgesia that persists after the return of sensation, during which time the need for strong analgesics is reduced. The half-life of Bupivacaine Hydrochloride in adults is 2.7 hours36. Bupivacaine was chosen for the purpose of this study since it is long-acting37 and likely to provide pain relief once the epidural analgesia has subsided.

   How will the information from the study be used? If the proposed hypothesis will be proven, better pain management could be offerred to women, and improve the quality of postpartum care. In addition, alleviation of postpartum perineal pain will enable women to take better care of their offspring.
2. The Proposed Trial

   2.1. Proposed Trial design

   The proposed trial will be a two-armed, randomized, single-masked, controlled trial

   2.2. Planned interventions

   2.2.1. Randomization

   Once a woman has consented to be considered for the trial, eligibility must be confirmed. Once eligibility has been confirmed, the women will be randomized into the study using computer-generated sequence and sealed envelopes to one of three study arms: Bupivacaine injection or sham injection to reflect current care.

   2.2.2. All study participants

   Prior to injection of the intervention drug, the patient will be asked to press the bolus button of the epidural analgesia; the time of this occurs will be recorded. The length of the 2PT/Epi will be measured in centimeters and documented. The laceration will be sutured using 2-0 Caprosyn suture. Subcuticular sutures will be used for skin closure.

   2.2.3. Bupivacaine arm

   The edges of the 2PT/Epi will be infiltrated with 10ml of Bupivacaine 0.5%+Epinephrine 50mcg prior to suture placement.

   2.2.4. Control arm

   Sham injection will be done using a syringe filled with 10ml of NaCl 0.9%, but the fluid will not be injected to the edges of the laceration but discarded. The sham injection will last no less than 10 seconds.

   2.3. Methods of protecting against bias

   The randomization will be done using a computer software. The patients and their companions will be asked not to observe the injection process. The physician performing the perineal repair will prepare the injection outside the patient's room. The nursing staff who will be directly involved with the care of the patients will be masked to the assigned arm.

   2.4. Planned inclusion/exclusion criteria

   2.4.1. Inclusion criteria
   * Maternal age > 18 years of age
   * Gestational age≥34 weeks of gestation
   * Vaginal delivery
   * Perineal laceration (2PT/Epi)
   * Effective epidural anesthesia
   * No known hypersensitivity to bupivacaine or amino-amide anesthetics

   2.4.2. Exclusion criteria
   * Medical history of a chronic pain syndrome
   * Intrapartum morphine use

   2.5. Duration of treatment period The treatment will be given as a single dose. Follow-up will take place for 24 hours after the last bolus dose.

   2.6. Primary outcome and other outcomes

   2.6.1. Primary outcome

   The primary outcome will be the proportion of women in the bupivacaine arm and the no analgesic arm who have a Numeric Rating Scale (NRS) score≤4 at 6-hours (±30 minutes) after last epidural bolus.

   Numeric Rating Scale (NRS)

   The NRS for pain is a unidimensional measure of pain intensity in adults. It is a segmented numeric version of the visual analog scale (VAS) in which a respondent selects a whole number (0-10 integers) that best reflects the intensity of their pain. The NRS is anchored by terms describing pain severity extremes, with 0 representing one pain extreme (e.g., "no pain") and 10 representing the other pain extreme (e.g., "pain as bad as you can imagine" and "worst pain imaginable"). The number that the respondent indicates on the scale to rate their pain intensity is recorded. Scores range from 0 -1013.

   Visual Analog Scale (VAS)

   The pain VAS is a continuous scale comprised of a horizontal or vertical line, usually 10 centimeters (100 mm) in length, anchored by 2 verbal descriptors, one for each symptom extreme. The respondent is asked to place a line perpendicular to the VAS line at the point that represents their pain intensity. The score is determined by measuring the distance (mm) on the 10-cm line between the "no pain" anchor and the patient's mark, providing a range of scores from 0-100 (mm) or 0-10 (cm). A higher score indicates greater pain intensity. Based on the distribution of pain VAS scores in postsurgical patients, the following cut points on the pain VAS have been recommended: no pain (0-4 mm), mild pain (5-44 mm), moderate pain (45-74 mm), and severe pain (75- 100 mm). No training is required other than the ability to use a ruler to measure distance to determine a score13.

   2.6.3. Other outcomes

   The following are the other outcomes which will be compared among the three intervention arms:
   * Time to first ambulation (getting out of bed).
   * Time to first analgesic administration.
   * Number of administration of additional analgesics in the first 24 hours after last epidural bolus.
   * NRS at 12 and 24 hours (±30 minutes) after last epidural bolus.
   * Highest NRS while in rest during the first 12 and 24 hours after last epidural bolus.
   * Highest NRS while sitting during the first 12 and 24 hours after last epidural bolus.
   * Highest NRS while walking during the first 12 and 24 hours after last epidural bolus.
   * Highest NRS while breastfeeding during the first 12 and 24 hours after last epidural bolus.

   2.7. Sample size and planned Recruitment Rate

   Group sample sizes of 323 in group one and 323 in group two achieve 80% power to detect a difference between the group proportions of -0.0990 (30% reduction). The proportion in group one (the treatment group) is assumed to be 0.3300 under the null hypothesis and 0.2310 under the alternative hypothesis. The proportion in group two (the control group) is 0.3300. The test statistic used is the two-sided Z test with pooled variance. The significance level of the test was targeted at 0.0500.

   To account for 10% loss to follow-up the sample size will be inflated to 355 per group. This will result in a total sample size of 710 for the 2 arms. The calculation was carried out using PASS Version 12 (Hintze, J. (2014). NCSS, LLC. Kaysville, Utah.).

   2.8. Analysis plan

   2.8.1. Interim Analysis

   An interim analysis of efficacy (the primary outcome) is planned when 50% of the total subjects have outcome data available. The group sequential method of Lan and DeMets will be used to characterize the rate at which the type I error is spent where the spending function is the O'Brien-Fleming boundary. The nominal alpha level at the interim analysis (50% of participants) is 0.0031 and at the final analysis (100%) is 0.049. In addition, a futility analysis will be conducted whereby the probability of finding a significant result at the end of the study will be calculated based on the current trend in the data, the null and alternative hypotheses.

   2.8.2. Final Analysis

   Descriptive statistics will be calculated for all variables of interest. Continuous measures such as age will be summarized using means and standard deviations whereas categorical measures will be summarized using counts and percentages.

   The primary outcome, proportion of women with NRS≥4 , will be compared between arms using tests of proportions.

   The secondary outcome, will be compared between arms using chi-square tests (or Fisher's exact tests in the case of low expected cell counts).

   The remaining outcome measures, such as Time to first ambulation, are continuous or interval measures. These will be assessed using t-tests or Wilcoxon rank sum tests in the case of non-normally distributed data.

   All analyses will be carried out using SAS Version 9.4 (SAS Institute, Cary, NC, USA).

ELIGIBILITY:
Inclusion Criteria:

* Maternal age > 18 years of age
* Gestational age≥34 weeks of gestation
* Vaginal delivery
* Perineal laceration (2PT/Epi)
* Effective epidural anesthesia
* No known hypersensitivity to bupivacaine or amino-amide anesthetics

Exclusion Criteria:

* Medical history of a chronic pain syndrome
* Intrapartum morphine use

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2018-09-14 (Actual); Primary Completion 2022-05-09 (Actual); Study Completion 2022-05-09 (Actual)

PRIMARY OUTCOMES:
Proportion of women who have a Numeric Rating Scale (NRS) score≤4 at 6-hours (±30 minutes) after last epidural bolus (comparison between bupivacaine arm and the no analgesic arm) | 6-hours (±30 minutes) after last epidural bolus.
  Comparison between the bupivacaine arm and the no analgesic arm in terms of pain score at 6-hours.

OTHER OUTCOMES:
Time to first ambulation (getting out of bed). | 24 hours
Number of administration of additional analgesics in the first 24 hours after last epidural bolus. | 24 hours
NRS (Numeric Rating Scale, 0-10, acceptable if < 3) at 12 and 24 hours (±30 minutes) after last epidural bolus | 12 and 24 hours
Highest NRS (Numeric Rating Scale, 0-10, acceptable if < 3) while in rest during the first 12 and 24 hours after last epidural bolus | 12 and 24 hours
Highest NRS (Numeric Rating Scale, 0-10, acceptable if < 3) while sitting during the first 12 and 24 hours after last epidural bolus | 12 and 24 hours
Highest NRS (Numeric Rating Scale, 0-10, acceptable if < 3) while walking during the first 12 and 24 hours after last epidural bolus | 12 and 24 hours
Highest NRS (Numeric Rating Scale, 0-10, acceptable if < 3) while breastfeeding during the first 12 and 24 hours after last epidural bolus | 12 and 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Amir Aviram, MD, Principal Investigator — Sunnybrook Health Sciences Centre
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided
Undecided yet.

REFERENCES:
- [Background] Khan GQ, Lilford RJ. Wound pain may be reduced by prior infiltration of the episiotomy site after delivery under epidural analgesia. Br J Obstet Gynaecol. 1987 Apr;94(4):341-4. doi: 10.1111/j.1471-0528.1987.tb03102.x. PMID 3580317
- [Background] Schinkel N, Colbus L, Soltner C, Parot-Schinkel E, Naar L, Fournie A, Granry JC, Beydon L. Perineal infiltration with lidocaine 1%, ropivacaine 0.75%, or placebo for episiotomy repair in parturients who received epidural labor analgesia: a double-blind randomized study. Int J Obstet Anesth. 2010 Jul;19(3):293-7. doi: 10.1016/j.ijoa.2009.11.005. Epub 2010 Jun 2. PMID 20627696